CLINICAL TRIAL: NCT06701149
Title: A Randomized, Open-label, Single-dose, Parallel Group Study to Compare the Pharmacokinetics of SIM0718 Injection in Healthy Adult Subjects in China
Brief Title: A Comparative Study of the Pharmacokinetics of SIM0718 Injection in Healthy Adult Subjects in China
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Simcere Pharmaceutical Co., Ltd (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: SIM0718-101
Record Dates: First submitted 2024-11-17; First posted 2024-11-22 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-11

CONDITIONS: Healthy Adult Subjects

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rademikibart injection (Experimental): Received subcutaneous injection administration on the morning of the first day .
  Interventions: Drug: Rademikibart injection
- CBP-201 injection (Active Comparator): Received subcutaneous injection administration on the morning of the first day.
  Interventions: Drug: CBP-201 injection

INTERVENTIONS:
Drug: Rademikibart injection — 300 mg administered subcutaneously on the first day
  Arms: Rademikibart injection
Drug: CBP-201 injection — 300 mg administered subcutaneously on the first day
  Arms: CBP-201 injection

SUMMARY:
A study to compare the pharmacokinetics, safety and immunogenicity of SIM0718 injection in healthy adult subjects in China

DETAILED DESCRIPTION:
This will be a single-center, open-label, single-dose, parallel group Comparative Study.

After meeting the eligibility criteria, all eligible participants will be randomized 1:1to an experimental group (Rademikibart injection) or an Active Comparator (CBP-201 injection) as defined in the protocol. Randomization will be stratified by protocol defined body weight categories.

The study will comprise:

A Screening Period up to 28 days. One treatment period during which eligible participants will be admitted to the Clinical Unit on Day-1 to reassess their eligibility. Participants who meet eligibility criteria will be randomized to receive 300mg subcutaneous (SC) of Rademikibart injection or CBP-201 injection on Day 1. Participants will be discharged on Day 8.

The participants will return to the center for Follow-up Visits on Days 10, 12, 15, 18, 22, 29, 36 43 and 57

ELIGIBILITY:
Inclusion Criteria:

* 1) Able to read, understand, and voluntarily sign the informed consent form.
* 2) Healthy adult male or female subjects aged 18~50 years (including the cut-off value) at screening.
* 3) The body mass index between 19 and 26 kg/m2 (including the cut-off value), and the weight of male subjects at least 50kg, and the weight of female subjects at least 45kg.
* 4) Subjects (including male subjects) and their spouses/partners have no pregnancy plan (including sperm donation and egg donation) for at least 90 days after signing the informed consent form to the last dose and voluntarily take effective non-drug contraceptive measures.
* 5)5) Able to communicate well with clinical staff and complete the trial in accordance with the protocol requirements.

Exclusion Criteria:

* 1) Subject has any clinically significant history of cardiovascular, respiratory (including asthma, bronchospasm), renal, hepatic, digestive, metabolic, endocrine, psychiatric, neurological, hematologic, or rheumatic disease, or has a psychiatric illness or disorder, or has a history of acute or chronic infections and other abnormalities that may affect safety or may affect the results of the study, as judged by the investigator.
* 2) Patients with severe infection or systemic infection within 8 weeks before administration, requiring intravenous anti-infection treatment or hospitalization due to infection; Those who have an infection (including chronic or local infection) within 7 days before administration; Those with a history of recurrent infections and underlying diseases that are prone to infection; Those who currently suffer from oral herpes or shingles.
* 3) Previous history of asthma, allergic reactions, allergic conjunctivitis, atopic dermatitis or other allergic diseases; History of significant allergy to any drug or previous serious adverse reaction to subcutaneous administration.
* 4) Known symptoms of dermatitis or skin abnormalities in and around the site of administration. The proposed injection site has skin depression, skin induration, scarring, inflammation, edema, ulcer, infection, bleeding and any other conditions that are not suitable for subcutaneous injection.
* 5) Those who have suffered from clinically significant major diseases or undergone major surgical operations within 1 month before dosing, or are expected to require major surgery during the trial.
* 6) Active tuberculosis, latent tuberculosis, or history of nontuberculous mycobacterial infection at screening Note:
* Unless there is a clear specialist document, evidence that the disease has been adequately treated, and biologics are currently acceptable (in the medical judgment of the investigator and/or infectious disease specialist);
* T-spot testing may be used to aid in the diagnosis of people with suspected tuberculosis, if needed.
* 7) Positive Treponema pallidum specific antibody (TP-Ab), hepatitis B surface antigen (HBsAg), hepatitis B core antibody (HBcAb), hepatitis C antibody (HCV-Ab), human immunodeficiency virus antigen/antibody (HIV Ag/Ab).
* 8) Abnormal vital signs at screening period or baseline as judged by the investigator to be clinically significant.
* 9) During the screening period, the laboratory examination was judged to be clinically significant by the investigator.
* 10) Female subjects who test positive for pregnancy during the screening period or baseline period or are lactating.
* 11) The 12-lead ECG showed QTcF ≥450 ms for males or QTcF ≥470 ms for females at screening, or there were other clinically significant ECG abnormalities, which the investigator judged to be inappropriate to participate in the study.
* 12) Use of prescription or over-the-counter drugs (including Chinese herbal medicines and health products) within 14 days or 5 half-lives (whichever is longer) before dosing.
* 13) Use of IL-4 drugs before screening, or treatment with biologics within 12 weeks or 5 half-lives (whichever is longer) prior to dosing.
* 14) Use of immunomodulatory drugs (including topical or systemic corticosteroids) within 4 weeks prior to the first dose.
* 15) Have received a live or live attenuated vaccine within 12 weeks prior to dosing, or will receive a live or live attenuated vaccine during the study or within 8 weeks after the last dose.
* 16) Participated in any clinical trial and received at least one trial administration within 3 months or 5 half-lives (whichever is longer) prior to dosing; Have donated blood or lost a large amount of blood (>400mL) within 3 months prior to dosing.
* 17) History of regular alcohol consumption, drinking more than 14 units of alcohol per week within 3 months prior to dosing (1 unit of alcohol = 285 mL of beer or 25 mL of spirits or 100 mL of wine); or have taken any alcohol-containing products within 48 hours before dosing; or those who have a positive alcohol breath test at the baseline visit.
* 18) Smoking more than 5 cigarettes or equivalent tobacco per day within 3 months before administration; History of drug abuse within the past five years or drug use within 3 months prior to dosing; or positive urine drug abuse screen at the screening visit/baseline visit.
* 19) Any other situation that the investigator believes may affect the subject's provision of informed consent or follow the trial protocol or judges that it is not suitable to participate in this trial, or the subject's participation in the trial may affect the trial results or their own safety.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 178 (Estimated)
Dates: Start 2024-11-28 (Estimated); Primary Completion 2025-02-28 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Primary pharmacokinetic (PK) parameters of SIM0718（Cmax） | Day0-Day57
  Primary pharmacokinetic (PK) parameters of a single subcutaneous administration of SIM0718 （Cmax）
Primary pharmacokinetic (PK) parameters of SIM0718（AUC0-t ） | Day0-Day57
  Primary pharmacokinetic (PK) parameters of a single subcutaneous administration of SIM0718 （AUC0-t ）
Primary pharmacokinetic (PK) parameters of SIM0718 （ AUC0-inf） | Day0-Day57
  Primary pharmacokinetic (PK) parameters of a single subcutaneous administration of SIM0718 （ AUC0-inf）

SECONDARY OUTCOMES:
Cmax of SIM0718 PK parameters | Day0-Day57
  including but not limited to Cmax
Adverse events of Safety of during the priod | Day（-28）-Day57
  Adverse events
The positive rate and titer of anti-drug antibodies of immunogenicity | Day0-Day57
  The positive rate and titer of anti-drug antibodies
AUC0-inf of SIM0718 PK parameters | Day0-Day57
  including but not limited to AUC0-inf
AUC0-t of SIM0718 PK parameters | Day0-Day57
  including but not limited to AUC0-t
AUC_%Extrap of SIM0718 PK parameters | Day0-Day57
  including but not limited to AUC_%Extrap
Tmax of SIM0718 PK parameters | Day0-Day57
  including but not limited to Tmax
t1/2 of SIM0718 PK parameters | Day0-Day57
  including but not limited to t1/2
CL/F of SIM0718 PK parameters | Day0-Day57
  including but not limited to CL/F
Vz/F of SIM0718 PK parameters | Day0-Day57
  including but not limited to Vz/F
λz of SIM0718 PK parameters | Day0-Day57
  including but not limited to λz
injection site reactions of Safety of during the priod | Day（-28）-Day57
  injection site reactions
vital signs of Safety of during the priod | Day（-28）-Day57
  vital signs (body temperature, pulse, blood pressure)
physical examination of Safety of during the priod | Day（-28）-Day57
  physical examination
12-lead electrocardiogram (ECG) of Safety of during the priod | Day（-28）-Day57
  12-lead electrocardiogram (ECG)
blood routine of Safety of during the priod | Day（-28）-Day57
  blood routine
urine routine of Safety of during the priod | Day（-28）-Day57
  urine routine
blood biochemistry of Safety of during the priod | Day（-28）-Day57
  blood biochemistry
coagulation function and other clinical laboratory examination indicators of Safety of during the priod | Day（-28）-Day57
  coagulation function and other clinical laboratory examination indicators
the positive rate of neutralizing antibodies of immunogenicity | Day0-Day57
  the positive rate of neutralizing antibodies
the effects of anti-drug antibodies of immunogenicity | Day0-Day57
  the effects of anti-drug antibodies
titers of immunogenicity | Day0-Day57
  titers
neutralizing antibodies on PK will be assessed if necessary of immunogenicity | Day0-Day57
  neutralizing antibodies on PK will be assessed if necessary

CONTACTS AND LOCATIONS:
Overall Officials: wen qing, Principal Investigator — Jinan Central Hospital